CLINICAL TRIAL: NCT02466464
Title: Use of Microporous Polysaccharide Hemospheres (MPH) in Management of Acute Epistaxis
Brief Title: Microporous Polysaccharide Hemospheres Epistaxis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients were successfully recruited
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Oswaldo A Henriquez, Principal Investigator, Emory University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB00070733
Record Dates: First submitted 2015-06-05; First posted 2015-06-09 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Epistaxis
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Microporous Polysaccharide Hemospheres (MPH) (Active Comparator): Subjects with acute epistaxis will receive microporous polysaccharide hemospheres (Arista) powder. In the event that Arista fails to assist in resolving nosebleed in 15 minutes, subjects will be promptly escalated to the control group and will receive Merocel.
  Interventions: Device: Microporous Polysaccharide Hemospheres; Device: Nasal Tampon
- Merocel (Control) (Active Comparator): Subjects with acute epistaxis will receive standard-of-care treatment, nasal tampon (Merocel). In the event that Merocel fails to assist in resolving nosebleed in 15 minutes, subjects will be promptly escalated to the MPH group and will receive Arista powder.
  Interventions: Device: Microporous Polysaccharide Hemospheres; Device: Nasal Tampon

INTERVENTIONS:
Device: Microporous Polysaccharide Hemospheres — Two grams of Arista powder will be placed into the nose followed by four minutes of pressure and a moustache dressing.
  Other Names: Arista
Device: Nasal Tampon — 8 cm of Merocel dressing will be placed into one or both sides of your nose for the next three to five days and will then be removed by the physician.
  Other Names: Merocel

SUMMARY:
The purpose of this study is to compare a new treatment for nosebleeds to the treatment that has been used for many years.

DETAILED DESCRIPTION:
Nosebleeds are a common condition which affect many Americans every day.The standard treatment in this hospital for nosebleeds that do not resolve with squeezing the nose or nasal spray is to place a nasal packing (aka nasal tampon) into the nose. This is an effective treatment in most cases, but patients may find it to be uncomfortable. The investigators will be comparing the standard nasal packing with a new type of powder which may also stop nosebleeds.

ELIGIBILITY:
Inclusion Criteria:

* acute epistaxis who have failed conservative measures (including application of pressure and application of oxymetazoline spray) and for which the Otolaryngology service has been consulted
* must be alert and oriented
* hemodynamically stable with a hemoglobin greater than 9 g/dL
* cooperative

Exclusion Criteria:

* unable to consent or cooperate
* history of hereditary hemorrhagic telengectasias
* hemophilia
* clotting factor deficiencies
* history of prior surgery for epistaxis control
* nasal trauma
* recent sinonasal surgery
* hemodynamic instability
* posterior bleed (as determined by Ear, Nose, Throat physician)
* visibly bleeding vessel
* allergy to product
* current diabetic ketoacidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Number of subjects with resolution of bleed | 15 minutes (average time to resolve bleeding)
  Resolution of bleeding is determined by cessation of blood flow anteriorly from the nares as well as posteriorly in the pharynx. This will be determined by the otolaryngology resident or attending managing the patient during the study.

SECONDARY OUTCOMES:
Time until resolution of bleeding | 15 minutes (average time to resolve bleeding)
  Number of minutes it takes to resolve bleeding comparing the Arista powder group versus the Merocel tampon group.

CONTACTS AND LOCATIONS:
Overall Officials: Oswaldo Henriquez Ajami, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Department of Otolaryngology Clinic, Atlanta, Georgia, United States